CLINICAL TRIAL: NCT03676569
Title: Intrathecal Autologous Adipose Derived Regenerative Cells Treatment of Autoimmune Determined Refractory Epilepsy - Evaluation of Safety and Efficacy
Brief Title: Intrathecal Autologous ADRC Treatment of Autoimmune Refractory Epilepsy
Acronym: EPIMSC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mossakowski Medical Research Centre Polish Academy of Sciences (Other)
Collaborators: Institute of Mother and Child, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Anna Sarnowska, M.D., Ph.D.; Head of Translative Platform for Regenerative Medicine MRC Mossakowski PAS, Mossakowski Medical Research Centre Polish Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17/2014 IMiD
Record Dates: First submitted 2018-09-14; First posted 2018-09-18 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Refractory Epilepsy
Keywords: autoimmune epilepsy; refractory epilepsy; ADRC; mezenchymal stem cells; anti-neuronal antibody; Rasmussen encephality; adipose derived regenerative stem cells
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: Experimental clinical treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Autologous ADRC transplantation in autoimmune refractory epilepsy
  Interventions: Biological: ADRC transplantation in autoimmune refractory epilepsy

INTERVENTIONS:
Biological: ADRC transplantation in autoimmune refractory epilepsy

SUMMARY:
Refractory epilepsies caused by an autoimmune mechanisms lead in children to progressive neurodegeneration. Immunomodulation therapy is effective only in a half of such cases. New approaches are undertaken. It was found that ADRC (adipose derived regenerative cells) isolated from adipose tissue consist mesenchymal stem cells that act as tissue repair cells. The purpose of this experimental study is to evaluate the possibility and safety of the use of multipotent mesenchymal adipose derived regenerative cells (ADRC) in patients diagnosed with an autoimmune determined refractory epilepsy.

Study protocol:

Intrathecal infusions of autologous ADRC obtained after liposuction followed by isolation by Cytori system will be performed. Procedure will be repeated 3 times every 3 months in each patient. Neurological status, brain MRI, cognitive function and antiepileptic effect will be supervised during 24 months.

DETAILED DESCRIPTION:
Epilepsy is a chronic neurological disorder diagnosed in about 1% of the population, or c. 400,000 patients in Poland. Autoimmune refractory epilepsy is rare but most disabled epilepsy leading to developmental regression. The belief in a positive effect of ADRCs in drug-resistant epilepsy comes from test results showing the ability of mesenchymal cells to concentrate in damaged tissues, as well as their strong immunomodulating, especially anti-inflammatory, properties. Patients with drug resistant epilepsy show decreased numbers of neurons within the epilepsy zone, with most of these being hyperactive and malfunctioning. Additionally, an inflammatory active reaction in affected brain tissue is visible. ADRC-induced activation of endogenous neurogenesis may increase chances that the epilepsy zone will be reduced, and give a positive impact as regards the neuropsychiatric disorders commonly present in patients with epilepsy. Another common process accompanying recurring epilepsy attacks is active inflammation. Per the literature, ADRCs show strong neuroprotective, immunomodulating and antiapoptotic qualities and they may potentially reduce the frequency of epilepsy attacks. Thus, a clinical trial with ADRCs, addressed to drug-resistant epilepsy sufferers would be promising in controlling the epileptic seizures and coexisting behavioral / psychiatric symptoms. The goal is to improve the quality of life of the patients and their caregivers.

In patients who were diagnosed with autoimmune drug-resistant epilepsy and have met the set criteria and qualified to take part in the examination, after a formal written consent of their parents at the Clinic of Child Neurology IMC neurological examination, routine laboratory tests, EEG and neuropsychological assessment will be performed. ADRC will be obtained after liposuction and isolation with Cytori system.

Before intrathecal transplantation of ADRC suspension ( 5 ml), cerebrospinal fluid will be collected for evaluation of origin protein level, oligoclonal bands, the IgG index as well as GluR3, VGKC complex/LGI1, GM1, NT-3, GAD, and NMDAR antibodies. At the same time there will be an intake of 5ml of serum to evaluate levels of immunoglobulins IgA, IgM and IgG.

Procedure will be repeated 3 times every 3 months in each patient. Neurological status, brain MRI, cognitive function and antiepileptic effect will be supervised during 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Drug-resistant epilepsy confirmed in anamnesis and diagnostic tests (EEG, MR)
* Children between 3 and 18 years old
* Presence of antineuronal antibody in serum or CSF
* Rasmussen encephalitis (proven cellular immunity pathogenesis)
* Probable autoimmune pathogenesis (autoimmune diseases in family, febrile infection associated refractory epilepsy)
* Willing and able to provide written informed consent (patient or legal guardian)

Exclusion Criteria:

* Refractory epilepsy with proven genetic or metabolic ethiology
* Neoplastic disease
* Active inflammatory process at the time of recruitment
* Coagulation disorder
* Status epilepticus
* Participation in another clinical trial
* Lack of willingness and ability to provide written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-11-15 (Actual); Primary Completion 2019-04-14 (Actual); Study Completion 2019-04-14 (Actual)

PRIMARY OUTCOMES:
Rate of epileptic seizures | 3 months
  recording of epileptic seizures frequency, EEG

SECONDARY OUTCOMES:
Intelligence test | 3 months
  The Leiter contains 10 subtests organized into four domains: Fluid Intelligence Visualization, Memory, Attention
School progress | 3 months
  teacher references

OTHER OUTCOMES:
Radiological assesment | 12 months
  MRI
The level of antineural antibodies | 3 months
  protein level, oligoclonal bands, IgG index as well as GluR3, VGKC complex/LGI1, GM1, NT-3, GAD, NMDAR antibodies from cerebrospinal fluid for evaluation the origin

CONTACTS AND LOCATIONS:
Overall Officials: Dorota Antczak-Marach, M.D., Principal Investigator — Institute of Mother and Child; Ewa Sawicka, Prof., Principal Investigator — Institute of Mother and Child

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Szczepanik E, Mierzewska H, Antczak-Marach D, Figiel-Dabrowska A, Terczynska I, Tryfon J, Krzesniak N, Noszczyk BH, Sawicka E, Domanska-Janik K, Sarnowska A. Intrathecal Infusion of Autologous Adipose-Derived Regenerative Cells in Autoimmune Refractory Epilepsy: Evaluation of Safety and Efficacy. Stem Cells Int. 2020 Jan 3;2020:7104243. doi: 10.1155/2020/7104243. eCollection 2020. PMID 32190059